CLINICAL TRIAL: NCT05267548
Title: A Prospective PMCF Study Investigating the Safety and Clinical Performance of the Oceanus 14pro, Oceanus 18 and Oceanus 35 Balloon Catheters, the Luminor 14m and Luminor 18 Drug Coated Balloons, the Angiolite BTK Sirolimus Eluting Peripheral Stent System and the Sergeant Peripheral Support Catheter for the Endovascular Intervention in Popliteal and Infrapopliteal Arteries
Brief Title: Investigating the Safety and Clinical Performance of Seven iVascular Devices for Endovascular Intervention in the Popliteal and/or Infrapopliteal Arteries
Acronym: POP-BTK
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: iVascular S.L.U. (Industry)
Collaborators: FCRE (Foundation for Cardiovascular Research and Education) (Other)
Responsible Party: Sponsor
Other Study IDs: FCRE-211206
Record Dates: First submitted 2022-02-24; First posted 2022-03-04 (Actual); Last update posted 2023-02-03 (Actual); Status verified 2023-02

CONDITIONS: Peripheral Arterial Disease Below The Knee

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No

SUMMARY:
The rationale of this study is to confirm and support the clinical safety and performance of the Oceanus 14pro, Oceanus 18 and Oceanus 35 Balloon Catheters, the Luminor 14m and Luminor 18 Drug Coated Balloons, the Angiolite BTK Sirolimus Eluting Peripheral Stent System and the Sergeant Peripheral Support Catheter in a real-word population of 143 patients who underwent an endovascular intervention the popliteal and/or infrapopliteal arteries within standard-of-care (SOC) where at least 1 of the investigational products from iVascular were used.

ELIGIBILITY:
Inclusion Criteria:

1. Corresponding to the CE-mark indications/contra-indications and according to the IFU of the device.
2. Patient is >18 years old.
3. Patient understands the nature of the procedure and provides written informed consent prior to enrolment in the study.
4. Target lesion(s) is/are located in the popliteal or infrapopliteal arteries
5. Patient is eligible for treatment with the Oceanus 14pro Balloon Catheter and/or the Oceanus 18 Balloon Catheter and/or the Oceanus 35 Balloon Catheter and/or the Luminor 14m DCB and/or the Luminor 18 DCB and/or the Angiolite BTK Sirolimus Eluting Peripheral Stent System and/or the Sergeant Peripheral Support Catheter as described in the IFU for each device.

Exclusion Criteria:

1. Anatomy or size of vessels that will not allow appropriate usage of the investigational devices, following IFU of the investigational devices.
2. Known contraindication and/or allergy to (a component of) an investigational device.
3. Pregnant women and women with childbearing potential not taking adequate contraceptives or currently breastfeeding.
4. Life expectancy of less than 12 months.
5. Any planned surgical intervention/procedure within 30 days after the study procedure.
6. Any patient considered to be hemodynamically unstable at onset of procedure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In this PMCF minimally invasive medical devices with special dedication towards the interventional cardiovascular field will be used. Indications for which the investigational devices are intended are listed in the protocol. Patients will be selected based on the investigator's assessment and evaluation of the underlying disease. The patient's medical condition should be stable, with no underlying medical condition which would prevent them from performing the required assessment or from completing the study. Patients should be geographically stable, willing and able to cooperate in this clinical study, and remain available follow-up.
Sampling Method: Non-Probability Sample
Enrollment: 143 (Estimated)
Dates: Start 2022-05-30 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Primary Safety Endpoint: Freedom from SAE/SADE | 2 years
  Freedom from Serious Adverse Events (SAEs) and Serious Adverse Device Effects (SADEs) during the procedure and up to 2 years after the procedure (depending on the device that was used).
Primary Efficacy Endpoint: Technical success | During procedure
  Technical success rate defined as successful crossing, introduction and deployment of the Oceanus 14pro Balloon Catheter and/or the Oceanus 18 Balloon Catheter and/or the Oceanus 35 Balloon Catheter and/or the Luminor 14m DCB and/or the Luminor 18 DCB and/or the Angiolite BTK Sirolimus Eluting Peripheral Stent System and/or the Sergeant Peripheral Support Catheter according to the respective IFU and without device related deficiencies.

SECONDARY OUTCOMES:
Physician Appraisal | During procedure
  General physician appraisal of the devices will be explored based on
  1. Simplicity of handling
  2. Pushability
  3. Trackability
  4. Crossability
  5. Profile Physician appraisal of the Luminor 14m and Luminor 18 Drug Coated Balloon Dilatation Catheters and the Oceanus 14pro, Oceanus 18 and Oceanus 35 Balloon Dilatation Catheters will be explored based on
  1. Deflation time 2. Balloon Compliance 3. Visibility 4. Balloon refolding Physician appraisal for the Angiolite BTK Sirolimus Eluting Peripheral Stent System will be explored based on
  1. Recoil
  2. Radial force
  3. Ease to canalize the lesion
  4. Stent coverage
  5. Stent graft recrossing
  6. Balloon refusal And physician appraisal for the Sergeant Peripheral Support Catheter will be explored based on
  1. Trackability over the guide wire 2. Absence of kinking behaviour 3. Injection Capacity 4. Ease of changing guide wires 5. Ease to canalize the lesion
Freedom from SAE | 2 years
  Freedom from SAE post-procedure and after 30 days, 1 year and 2 years (depending on the device that was used)
Freedom from SADE | 2 years
  Freedom from SADE post-procedure and after 30 days, 1 year and 2 years (depending on the device that was used)
Freedom from TLR | 2 years
  Freedom from Target Lesion Revascularization post-procedure and after 30 days, 1 year and 2 years (depending on the device that was used), defined as freedom from a repeat intervention to maintain or re-establish patency within the region of the treated arterial vessel plus 5mm proximal and distal to the treated lesion edge.

CONTACTS AND LOCATIONS:
Locations (8):
- Belgium (8):
  - Imelda Bonheiden, Bonheiden
  - Jessa Hasselt, Hasselt
  - Az Groeninge Kortrijk, Kortrijk
  - Az Sint Maarten Mechelen, Mechelen
  - HH Mol, Mol
  - Az Damiaan Oostende, Ostend
  - RZ Tienen, Tienen
  - Az Jan Portaels Vilvoorde, Vilvoorde

IPD SHARING:
Plan to Share IPD: No